CLINICAL TRIAL: NCT00873496
Title: Effects of Hydroxychloroquine on Oral Complaints of Sjögren Patients: a Prospective Sample Study.
Brief Title: Effects of Hydroxychloroquine on Oral Complaints of Sjögren Patients
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Esin Alpoz, Ege University School of Dentistry
Other Study IDs: EAlpoz 1
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Sjögren's Syndrome; Xerostomia
Keywords: Sjögren's Syndrome; hyposalivation; mouth dryness; complications
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia | interventions — Hydroxychloroquine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sjögren: Pre and post treatment establishment of salivary flow rate, objective and subjective clinical oral complications' severity of the patients using hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine

SUMMARY:
Chronic inflammation that comprises the exocrine glands' function leads to xerophthalmia and xerostomia in Sjögren's syndrome. The oral consequences range widely and they are related to decreased salivary output. Hydroxychloroquine may inhibit cholinesterase activity in salivary glands via interference with antigen processing mechanism, and thus, the investigators' hypothesis was that salivary gland function may be improved if treated with hydroxychloroquine. The effects of hydroxychloroquine on the salivary flow rate, subjective and objective parameters of the patients were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were recently diagnosed with primary SS according to American-European criteria and who were scheduled for HCQ treatment in Ege University Faculty of Medicine, Department of Rheumatology

Exclusion Criteria:

* Sjögren patients consuming alcohol or tobacco

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study group consisted of 30 female patients recently diagnosed as Sjögren's syndrome.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Salivary flow rate, objective and subjective clinical oral complaints | 2005 Jan-2009 Jan

CONTACTS AND LOCATIONS:
Overall Officials: Esin Alpoz, Study Director — Ege University School of Dentistry
Locations (1):
- Ege University School of Dentistry, Izmir, Bornova, Turkey (Türkiye)

REFERENCES:
- [Background] Alpoz E, Guneri P, Onder G, Cankaya H, Kabasakal Y, Kose T. The efficacy of Xialine in patients with Sjogren's syndrome: a single-blind, cross-over study. Clin Oral Investig. 2008 Jun;12(2):165-72. doi: 10.1007/s00784-007-0159-3. Epub 2007 Nov 14. PMID 18000691
- [Result] Kruize AA, Hene RJ, Kallenberg CG, van Bijsterveld OP, van der Heide A, Kater L, Bijlsma JW. Hydroxychloroquine treatment for primary Sjogren's syndrome: a two year double blind crossover trial. Ann Rheum Dis. 1993 May;52(5):360-4. doi: 10.1136/ard.52.5.360. PMID 8323383
- [Result] Dawson LJ, Caulfield VL, Stanbury JB, Field AE, Christmas SE, Smith PM. Hydroxychloroquine therapy in patients with primary Sjogren's syndrome may improve salivary gland hypofunction by inhibition of glandular cholinesterase. Rheumatology (Oxford). 2005 Apr;44(4):449-55. doi: 10.1093/rheumatology/keh506. Epub 2004 Dec 8. PMID 15590764